CLINICAL TRIAL: NCT02943759
Title: Resolution of Pain and Swelling After the Use of Neem Leaf Extract (Azadirachta Indica) Compared to Chlorhexidine Gluconate as an Intracanal Irrigant in Necrotic Primary Molar Teeth in Children Undergoing Pulpectomy Treatment: A Randomised Controlled Trial
Brief Title: Resolution of Pain and Swelling After the Use of Neem Leaf Extract Compared to Chlorhexidine Gluconate as an Intracanal Irrigant During Pulpectomy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mennatallah Sameh Ahmed Farouk Abdelhamid, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Chx_neemleaf
Record Dates: First submitted 2016-10-21; First posted 2016-10-25 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Periapical Abscess
MeSH Terms: conditions — Periapical Abscess | interventions — chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neem leaf extract (Experimental): Neem leaf extract (alcoholic solution) used as an anti inflammatory , antibacterial irrigant
  Interventions: Drug: Neem leaf extract
- Chlorhexidine gluconate (Active Comparator): 2% chlorhexidine gluconate intracanal irrigant solution used as an antibacterial chemical mean for canal irrigation
  Interventions: Drug: Chlorhexidine gluconate

INTERVENTIONS:
Drug: Neem leaf extract — A natural irrigant solution act as anti-inflammatory and anti bacterial
  Arms: Neem leaf extract
Drug: Chlorhexidine gluconate — 2%chlorhexidine gluconate , anti bacterial root canal irrigant solution
  Other Names: Gluconate-Chex 2%
  Arms: Chlorhexidine gluconate

SUMMARY:
The trial is to test the resolution of pain, swelling and other signs of periapical infection and the antimicrobial efficacy when using the neem leaf extract compared to chlorhexidine as root canal irrigant in Pulpectomy treatment for children.

DETAILED DESCRIPTION:
To compare the effectiveness of neem leaf extract with that of Chlorhexidine gluconate when used as an intracanal irrigant in primary molar teeth indicated for pulpectomy treatment.

P: children with primary necrotic molars indicated for pulpectomy I: Neem leaf extract (alcoholic solution). C: 2% chlorhexidine gluconate. O: Pain and swelling resolution. T:Over 12 months. S: Randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient and parent cooperation.

  * Absence of any systemic disease that would contraindicate pulp therapy.
  * Non vital molar teeth presenting with an acute or chronic periapical infection as a result of pulp necrosis ( Periapical abscess ,a sinus tract formation as a sequelae )
  * Making sure the patient is not taking an antibiotic and has not taken it for the past 2 weeks.
  * Absence of physiologic or pathologic root resorption that contraindicate pulp therapy.
  * Restorable teeth
  * Molars with at least two thirds of root remaining.

Exclusion Criteria:

* Children with any condition that contraindicates pulp therapy will be excluded (rheumatic fever, infective endocarditis , leukemia , corticosteroid therapy and immunosuppressed children).

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Pain | 1 year
  Patient reported pain and pain on percussion , binary
Swelling | 1 year
  Visual examination ,binary
Mobility | 1 year
  Mobility test ,binary

SECONDARY OUTCOMES:
Bacterial load | 48 hours
  Bacteria on culture plates measuring unit CFU/ml
Periapical pathosis | 1 year
  Periapical radiograph , binary

CONTACTS AND LOCATIONS:
Overall Officials: Dalia M Moheb, Assoc Prof, Study Director — Pediatric Dentistry & Dental Public Health Faculty of Oral & Dental Medicine , Cairo university; Norhan A El Dokky, Assoc Prof, Study Director — Pediatric Dentistry & Dental Public Health Faculty of Oral & Dental Medicine , Cairo university
Locations (1):
- Pediatric dentistry and Public health department-Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dutta A, Kundabala M. Comparative anti-microbial efficacy of Azadirachta indica irrigant with standard endodontic irrigants: A preliminary study. J Conserv Dent. 2014 Mar;17(2):133-7. doi: 10.4103/0972-0707.128047. PMID 24778508
- [Background] Ercan E, Ozekinci T, Atakul F, Gul K. Antibacterial activity of 2% chlorhexidine gluconate and 5.25% sodium hypochlorite in infected root canal: in vivo study. J Endod. 2004 Feb;30(2):84-7. doi: 10.1097/00004770-200402000-00005. PMID 14977302
- [Background] Louwakul P, Prucksathamrongkul W. The effect of 2% chlorhexidine as root canal irrigant in pulpectomies of primary molars. Pediatr Dent. 2012 Nov-Dec;34(7):e192-6. PMID 23265154
- [Background] Podar R, Kulkarni GP, Dadu SS, Singh S, Singh SH. In vivo antimicrobial efficacy of 6% Morinda citrifolia, Azadirachta indica, and 3% sodium hypochlorite as root canal irrigants. Eur J Dent. 2015 Oct-Dec;9(4):529-534. doi: 10.4103/1305-7456.172615. PMID 26929692
- [Background] Ruiz-Esparza CL, Garrocho-Rangel A, Gonzalez-Amaro AM, Flores-Reyes H, Pozos-Guillen AJ. Reduction in bacterial loading using 2% chlorhexidine gluconate as an irrigant in pulpectomized primary teeth: a preliminary report. J Clin Pediatr Dent. 2011 Spring;35(3):265-70. doi: 10.17796/jcpd.35.3.y052311j23617837. PMID 21678668